CLINICAL TRIAL: NCT05886543
Title: Pilates Exercise and Lung Functions in Postburn Inhalation Injury Patients.
Brief Title: Pilates Exercise and Inhalation Injury Post Burn
Acronym: burn
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Khadra Mohamed Ali (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, Khadra Mohamed Ali, assisst professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 341989
Record Dates: First submitted 2023-05-15; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Inhalation Injury
Keywords: Pilates exercise ,lung functions ,inhalation injury
MeSH Terms: interventions — Exercise Movement Techniques

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control group (Experimental): this group includes 30 patients who have post burn inhalation injury will receive conventional chest physiotherapy for(15-20) minutes 3times/week and medical treatment for 4 weeks as a total period of treatment.
  • computerized spirometer assessment before treatment are ( The following variables were measured: forced vital capacity (PVC%) and forced ·expiratory volume in one second (FEVl %) and peak expiratory flow (PEF %)and after one month
  Interventions: Behavioral: Conventional chest physical therapy; Behavioral: Pilates exercise
- study group (Experimental): this group includes 30 patients who have post burn inhalation injury will receive pilates exercise in addition to their conventional chest physiotherapy for(15-20) minutes 3times/week and medical treatment for 4 weeks as a total period of treatment.omputerized spirometer assessment before treatment are ( The following variables were measured: forced vital capacity (PVC%) and forced ·expiratory volume in one second (FEVl %) and peak expiratory flow (PEF %)and after one month
  Interventions: Behavioral: Conventional chest physical therapy; Behavioral: Pilates exercise

INTERVENTIONS:
Behavioral: Conventional chest physical therapy — Conventional chest physical therapy: The patients performed four series of five breath with 3 seconds of sustained breathing interspersed with periods of quite breathing followed by two or three coughs or huffs (with wound support by a pillow or his/her hands), twice a day in the first two postburned days and once a day from the third to the tenth days.
Behavioral: Pilates exercise — The Pilates technique, which stretched laterally and to the back, stressed costal breathing, in which the ribs climb and drop throughout the ventilatory stream. The transverse muscle had to work harder to avoid abdominal distension, provide more support to the diaphragm to promote lower rib movement, and provide more diaphragmatic excursion, During the expiratory phase, the transversus abdominis, the multifidus and the pelvic floor musculature were contracted.

SUMMARY:
Sixty patients with 25-45 years of age presenting post burn inhalation injury, randomly distributed into two equal groups, 30 patients for each group. control group receive conventional chest physiotherapy (diaphragmatic respiratory exercises, apical breathing exercises) for (15-20) minutes 3times/week and medical treatment for 4 weeks as a total period of treatment. study group will receive pilates exercise in addition to their conventional chest physiotherapy for (15-20) minutes 3times/week and medical treatment for 4 weeks as a total period of treatment, computerized spirometer assessment before treatment are ( The following variables were measured: forced vital capacity (PVC%) and forced ·expiratory volume in one second (FEVl %) and peak expiratory flow (PEF %)and after one month

DETAILED DESCRIPTION:
Two groups of sixty patients (thirty patients in each group) of both sexes of inhalation injury post burn are selected randomly to participate in the study.

The patients will be divided into two equal groups in number:

* Group (A) study group: this group includes 30 patients who have postburn inhalation injury will receive conventional chest physiotherapy (diaphragmatic respiratory exercises, deep inhalation exercises, and respiratory exercises associated with shoulder flexion movements and extension of the upper limbs, assisted cough, circulatory exercises and early ambulation) and medical treatment and pilates method.
* Group (B) control group: this group includes 30 patients who have postburn inhalation injury will receive conventional chest physiotherapy (diaphragmatic respiratory exercises, deep inhalation exercises, and respiratory exercises associated with shoulder flexion movements and extension of the upper limbs, assisted cough, circulatory exercises and early ambulation) and medical treatment.
* computerized spirometer assessment before treatment are ( The following variables were measured: forced vital capacity (PVC%) and forced ·expiratory volume in one second (FEVl %) and peak expiratory flow (PEF %)and after one month

ELIGIBILITY:
Inclusion Criteria:

* Age ranged between 25-45 years.
* All patients presented post-burn inhalation injury.
* Patients with facial burn or upper limb burn.
* All patients would be free of acute or chronic pulmonary disease and will have the capacity to perform the protocol evaluation tests properly.
* All patients enrolled to the study would have their informed consent.

Exclusion Criteria:

* Cardiac diseases.
* Chronic pulmonary disorders.
* Previous or present smoking history.
* Female patients who are pregnant and lactating.
* Post-burn patient on ICU.

Ages: 25 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2021-09-30 (Actual); Primary Completion 2021-11-20 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Measurement of Pulmonary Function (spirometry) | one month
  Spirometric evaluation had been undertaken on pre-rehabilitation. The following variables were measured: forced vital capacity (PVC%) and forced ·expiratory volume in one second (FEVl %) and peak expiratory flow (PEF %), by spirometry (ZAN 100 Handy 11- TB 100 E006) with the subject upright sitting or lying in the supine posture

SECONDARY OUTCOMES:
Measurement of anthropometric parameters. | before spirometer test
  Before spirometry testing, height and weight should be determined to find the body mass index essential in spirometry test. Standing height was measured in centimeters with· a measuring scale. Weight was measured in kilograms on a standardized weighing machine

CONTACTS AND LOCATIONS:
Overall Officials: Ali, a, Principal Investigator — assist professor - department of physical therapy for surgery - Cairo university
Locations (1):
- faculty of physical therapy , Cairo university, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No